CLINICAL TRIAL: NCT06222125
Title: A Phase II, Open-Label, Multicenter Study to Evaluate the Safety and Efficacy of HB0025 in Patients With Advanced Renal Cancer
Brief Title: A Study of HB0025 Injection in Patients With Advanced Renal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huabo Biopharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HB0025-0101
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Renal Cancer
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Intervention Model Description: Sequential Assignment This study will enroll 20 subjects at 10mg/kg and 20mg/kg respectively every 2 weeks (Q2W)to compare the safety and efficacy, and will be extended to the group with better efficacy and tolerance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): 10 mg/kg intravenously, every 2 weeks, till tumor progression or intolerance.
  Interventions: Drug: HB0025
- Arm 2 (Experimental): 20 mg/kg intravenously, every 2 weeks, till tumor progression or intolerance.
  Interventions: Drug: HB0025

INTERVENTIONS:
Drug: HB0025 — HB0025 IV every 2 weeks (q2w)
  Other Names: Recombinant humanized anti-programmed cell death-ligand 1（Anti-PD-L1） monoclonal antibody-VEGFR1 fusion protein

SUMMARY:
It is a phase II open label, multicenter study to assess the safety, tolerability, pharmacokinetics, and efficacy of HB0025 in patients with advanced clear cell renal cell carcinoma (ccRCC).

DETAILED DESCRIPTION:
The phase II study will enroll subjects with advanced clear cell renal cell carcinoma (ccRCC) who have progressing tumor after standard therapy and have no better treatment option.This study will set up 2 dose groups.HB0025 injection is administered once every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female. Age ≥ 18 years.
* The subject is able to understand and willing to sign the informed consent form (ICF) ; willing and able to comply with all study procedures.
* Patients with histologically and/or cytologically confirmed advanced clear cell renal cell carcinoma (defined as more than 50% clear cell component) that is not suitable for radical treatment or recurrence / metastasis, with or without sarcomatoid features; may benefit from investigational drug therapy as judged by the investigator; and who have disease progression after receiving at least one previous systemic treatment regimen (tyrosine kinase drugs such as sunitinib, axitinib, pazopanib, sorafenib, etc., other drugs such as everolimus, excluding treatment with immune checkpoint inhibitors) or who cannot tolerate the current standard treatment as judged by the investigator.
* At least one measurable tumor lesion was present according to RECIST 1.1. At the same scan level of CT or MRI scan, the longest diameter of non-lymph node lesions is at least 10 mm, and the short diameter of lymph node lesions is ≥ 15 mm. A baseline imaging assessment could be performed up to 28 days before the first dose.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1.
* Life expectancy ≥3 mouths
* liver function requirements:

  1. Total bilirubin (TBIL) ≤ 1.5×ULN
  2. Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5×ULN; AST or ALT ≤5×ULN if liver metastases are present.
* Creatinine (Scr) < 1.5×ULN and Calculated creatinine clearance (CrCL) > 40 mL/ min (Cockcroft-Gault Equation).
* Hematology：

  1. absolute neutrophil count (ANC) ≥ 1,500/µL. (No use of recombinant human granulocyte colony-stimulating factor to support treatment within 14 days before the first administration of HB0025).
  2. hemoglobin (HGB) ≥ 9 g/dL. (No transfusion or hemoglobin support within 14 days of HB0025 first administration).
  3. platelets (PLT) ≥ 75,000/µL. (No transfusion or recombinant human thrombopoietin support within 14 days of HB0025 first administration).

Exclusion Criteria:

* Have clinically active central nervous system (CNS) metastases. Patients with asymptomatic brain metastases who have been in a stable condition of imaging and neurological evaluation for more than 4 weeks after receiving relevant treatment will be allowed. Patients who have undergone hormone therapy can be enrolled only if the hormone therapy dose is less than 10 mg/day prednisone or the equivalent dose of other hormones for at least 2 weeks.
* Active autoimmune disease or history of autoimmune disease requiring systemic therapy < 2 years prior to screening except hypothyroidism, vitiligo, Grave's disease, Hashimoto's disease, or Type I diabetes. Patients with childhood asthma or atopy that has not been active in the 2 years prior to study screening are eligible.
* History of Grade 3-4 immune-related adverse events (irAEs) or irAEs requiring discontinuation of prior therapies, (except for grade 3 endocrinopathy that is managed with hormone replacement therapy).
* Use of systemic corticosteroids in a dose equivalent to >10 mg/day of prednisone or other immunosuppressive agent < 2 weeks prior to screening; the use of topical, intraocular, intraarticular, intranasal, or inhaled corticosteroids and systemic steroids to prevent (e.g., allergy to contrast agents) or treat non-autoimmune condition (e.g., delayed hypersensitivity caused by exposure to allergens) will be allowed.
* Cerebrovascular accident (CVA), transient ischemic attack (TIA), myocardial infarction (MI), unstable angina, or New York Heart Association (NYHA) class III or IV heart failure < 6 months of study entry; uncontrolled arrhythmia < 3 months of study entry; mean ECG QT-interval corrected according to Fridericia's formula (QTcF) > 470 milliseconds (ms) (male) or QTcF > 480 ms (female) obtained from three ECGs.
* Uncontrolled diabetes, glycosylated hemoglobin HbA1c >8%；
* Those who have previously received PD-1 pathway inhibitors or cytotoxic T lymphocyte associated antigen-4 (CTLA-4) antibodies or macromolecular vascular endothelial growth factor (VEGF) inhibitors (such as bevacizumab, ramucirumab, etc.).
* Anticancer therapy or radiation < 5 half-lives or 4 weeks (whichever is shorter) prior to study entry; palliative radiotherapy to a single area < 2 weeks prior to study screening is permitted. Measurable lesions cannot be previously irradiated unless they have demonstrated growth after radiation therapy (According to RECIST v1.1).
* Patients who have previously received allogeneic stem cell, Bone marrow or solid organ transplantation.
* Concurrent malignancy < 5 years prior to entry other than adequately treated cervical carcinoma-in-situ, localized squamous cell cancer of the skin, basal cell carcinoma, localized prostate cancer, ductal carcinoma in situ of the breast, or < T1 urothelial carcinoma.
* Any of the following infections:

  1. Active infection unresolved less than 2 weeks prior to first dose of study drug.
  2. Active Pulmonary tuberculosis.
  3. Positive results for HIV test.
  4. Active hepatitis B or C. Patients with asymptomatic hepatitis B virus carriers (HBV DNA titer < 1000 cps/mL or 200 IU/mL) or cured hepatitis C (negative hepatitis C virus RNA test) can be enrolled.
* Major surgery < 4 weeks prior to the first dose; Minor surgery < 2 weeks prior to the first dose.
* History of severe allergic reactions, grade 3-4 allergic reactions to treatment with another monoclonal antibody or known to be allergic to protein drugs or recombinant proteins or excipients in HB0025 drug formulation.
* Have received or will receive a live vaccine within 30 days prior to the screening.
* Pregnant or breastfeeding women.
* Patients who have participated in any clinical trial of a drug or medical device within 30 days prior to the first dose or participate in other drug clinical trials, the elution period of the test drug has not reached 5 half-lives.
* Any other serious underlying medical condition (e.g., active gastric ulcer, uncontrolled seizures, cerebrovascular incidents, gastrointestinal bleeding, severe signs and symptoms of coagulation and clotting disorders, cardiac conditions), or psychiatric, psychological, familial condition or geographical location that, in the judgment of the Investigator, may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment.
* Fertile subjects who do not want to use effective contraception during HB0025 treatment and within 90 days after the last dose.
* Positive COVID-19 quantitative real time (qRT) polymerase chain reaction (PCR) or rapid screening test during screening, except for patients who turned negative 1 week before administration without comorbidities and required more than 2 negative tests at intervals of not less than 72 hours.
* Patients with a history of arterial or deep vein thrombosis within 6 months before enrollment; evidence or history of a bleeding tendency within 2 months before enrollment.
* Severe dyspnea, pulmonary insufficiency or the need for continuous supportive oxygen therapy.
* Unhealed wound or ulcer; fractures from any cause within 3 months before screening
* Conditions that may cause bleeding or perforation of the digestive tract (such as duodenal ulcer, intestinal obstruction, Crohn's disease, Ulcerative colitis, large gastrectomy and small bowel resection, etc.); Patients with a history of intestinal perforation and fistula, who were not cured after surgical treatment; Esophageal and gastric varices.
* Immunomodulators, including but not limited to cyclosporine and tacrolimus, were administered within 2 weeks before enrollment.
* Other conditions which would make it inappropriate for the patient to participate as judged by the investigator.
* Arterial hypertension (systolic blood pressure > 140 mmHg or diastolic blood pressure ≥ 100 mmHg) that could not be controlled even with standard treatment.
* Patients with urine protein ≥ 2 + using test strips should have 24-hour urine collection, and patients with 24-hour urine protein content ≥ 2g.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 24 mouths
  ORR defined as the number of patients were confirmed complete response(CR) and/or partial response(PR) according to RECIST 1.1 divided by the patients with at least one tumour evaluation.

SECONDARY OUTCOMES:
Disease control rate (DCR) | up to 24 mouths
  DCR defined as the number of patients were confirmed CR and/or PR and/or stable disease(SD) according to RECIST 1.1 divided by the patients with at least one tumour evaluation
Progression-free Survival（PFS） | up to 24 mouths
  progression-free survival (PFS) means the time between the start of treatment and the onset of tumor progression or death from various causes.
Duration of response (DOR) | up to 24 mouths
  DOR defined as time from the first record of CR or PR to the first record of tumor progression or death of subjects
AUC | up to 24 mouths
  Area Under concentration-time Curve (AUC)
Cmax | up to 24 mouths
  Maximum serum concentration (Cmax)
Tmax | up to 24 mouths
  half-life time of maximum concentration
Anti-drug antibody (ADA) | up to 24 mouths
  Using the ELISA method to detect the anti-drug antibody production in peripheral blood after HB0025 administration.
Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) | up to 24 mouths
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Number of Participants With Abnormal Laboratory Parameters Reported as TEAEs | up to 24 mouths
  Participants with abnormal laboratory parameters reported as TEAEs are reported. Laboratory analysis included hematology, clinical chemistry, thyroid function tests, and urinalysis.
Number of Participants With Abnormal Vital Signs and Physical Examination Reported as TEAEs | up to 24 mouths
  Participants with abnormal vital signs (heart rate, blood pressure, temperature, and respiratory rate) and physical examination reported as TEAEs are reported.
Number of Participants With Notable QTc Interval | up to 24 mouths
  Notable QTc intervals included single beat changes from baseline (Day 1) values (> 30, > 60, and > 90 milliseconds). Participants who had notable QTc interval are reported.

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, MD/PHD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No